CLINICAL TRIAL: NCT02375958
Title: A Phase 1 Multi-center, Open-label Dose Escalation and Expansion Study of PCA062 Administered Intravenously in Adult Patients With p-CAD Positive Tumors
Brief Title: PCA062 in pCAD-positive Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPCA062X2101; 2014-003732-40 (EudraCT Number)
Record Dates: First submitted 2015-02-09; First posted 2015-03-03 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-02

CONDITIONS: Triple Negative Breast Cancer; Head & Neck Cancer; Esophageal Cancer
Keywords: PCA062; Triple Negative Breast Cancer; Head & Neck Cancer; Esophageal Cancer; pCAD, pcadherin, solid-tumors
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Head and Neck Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Triple Negative Breast Cancer (Experimental)
  Interventions: Drug: PCA062
- Head and Neck Cancer (Experimental)
  Interventions: Drug: PCA062
- Esophageal Cancer (Experimental)
  Interventions: Drug: PCA062

INTERVENTIONS:
Drug: PCA062

SUMMARY:
A first-in-human sttudy using PCA062 in patients with p-CAD positive solid tumors.

ELIGIBILITY:
Inclusion criteria:

1. Male or female ≥ 18 years of age
2. Documented pCAD expressing tumor cells with the exception of HNSCC and ESCC. An archived tumor sample collected within 36 months prior to baseline if available, or a new tumor biopsy sample must be available for molecular pre-screening.
3. Consent for a tumor biopsy at screening
4. Progressive disease and no effective therapy exists
5. Measurable disease as per RECIST v1.1 criteria
6. ECOG Performance status of ≤ 2

Exclusion criteria:

1. CNS metastatic involvement
2. Clinically significant cardiac, respiratory, gastrointestinal, renal, hepatic or neurological conditions.
3. A history of serious allergic reactions, which in the opinion of the investigator pose an increased risk of serious infusion reactions.
4. Monocular vision or has media opacities or any other condition that precludes monitoring of the retina or the fundus, or has a history of ophthalmology exam with retina or cornea abnormalities
5. Previously treated with anti-pCAD biologic therapies.
6. Received anti-cancer therapies within the following time frames prior to the first dose of study treatment:

   * Conventional cytotoxic chemotherapy: ≤4 weeks
   * Biologic therapy (eg, antibodies), other than ADCs: ≤4 weeks
   * Non-cytotoxic small molecule therapeutics: ≤5 T1/2 or ≤2 weeks (whichever is longer)
   * Other investigational agents: ≤4 weeks
   * Radiation therapy (palliative setting is allowed.): ≤4 weeks
   * Major surgery: ≤2 weeks
7. Patient has out of range laboratory values defined as:

   * Hematological values:
   * Absolute neutrophil count (ANC) <1.5 x 109/L
   * Hemoglobin (Hgb) <9 g/dL
   * Platelets <100 x 109/L
   * Hepatic and renal function
   * Total bilirubin >1.5 x upper limit of normal (ULN). For patients with Gilbert's syndrome, total bilirubin >2.5 x ULN.
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 x ULN for patients without tumor involvement of the liver or >5 x ULN for patients with tumor involvement of the liver.
   * Serum creatinine >1.5 x ULN and/or measured creatinine clearance < 40 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose limiting toxicities | 28 days

SECONDARY OUTCOMES:
Incidence and severity of serious/adverse events | Duration of study (each treatment cycle = 14 days)
Pharmacokinetic parameter Cmax | 84 days
  Cmax = the maximum concentration (peak) of the drug observed in the blood after a single administration of the drug
Presence of PCA062 anti-bodies | 84 days
  The presence and/or concentration of the anti-bodies will be tested from the blood samples collected
Overall response rate | Duration of study (each treatment cycle = 14 days)
Duration of response | Duration of study (each treatment cycle = 14 days)
Progression free survival | 18 months
Disease control rate | 18 months
Best overall response | Duration of study (each treatment cycle = 14 days)
Pharmacokinetic paramater Tmax | 84 days
  Tmax = the time the drug takes to reach maximum (peak) concentration in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (2):
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
- Novartis Investigative Site, Villejuif, France
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Koto Ku, Tokyo, Japan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duca M, Lim DW, Subbiah V, Takahashi S, Sarantopoulos J, Varga A, D'Alessio JA, Abrams T, Sheng Q, Tan EY, Rosa MS, Gonzalez-Maffe J, Sand-Dejmek J, Fabre C, Martin M. A First-in-Human, Phase I, Multicenter, Open-Label, Dose-Escalation Study of PCA062: An Antibody-Drug Conjugate Targeting P-Cadherin, in Patients With Solid Tumors. Mol Cancer Ther. 2022 Apr 1;21(4):625-634. doi: 10.1158/1535-7163.MCT-21-0652. PMID 35131875
- See also: Results for CPCA062X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17441